CLINICAL TRIAL: NCT05473247
Title: The Adaption of the GameSquad Exergaming Intervention for Young Adults With Down Syndrome: A Pilot Feasibility Study
Brief Title: GameSquad for Adults With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kameron Suire, Postdoctoral Researcher, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00148828
Record Dates: First submitted 2022-07-13; First posted 2022-07-25 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Down Syndrome; Physical Inactivity
MeSH Terms: conditions — Down Syndrome; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ring-Fit Adventure Group (Experimental): In Phase 1, participants will be asked to play Ring-Fit Adventure for 60 minutes per week for 4 weeks. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  In Phase 2, participants will be asked to play Ring-Fit Adventure for 60 (wk 1), 90 (wk 2), 120 (wk 3), and 150 (wk 4-12) minutes per week. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  Interventions: Behavioral: Ring-Fit Adventure Group

INTERVENTIONS:
Behavioral: Ring-Fit Adventure Group — Participants will be asked to play the exergame software, Ring-Fit Adventure, and attend weekly virtual health coaching sessions.

SUMMARY:
The investigators are assessing acceptability, appropriateness, and feasibility of the adapted GameSquad-DS intervention using validated scales alongside qualitative data among young adults with Down Syndrome. Specifically, the investigators will assess mins/wk of Ring-Fit Adventure played, attendance at 30 min. virtual health coaching sessions, semi-structured interviews, participant retention, and intervention safety measured as number of adverse events.

DETAILED DESCRIPTION:
Adults with DS face unique barriers to participation in MVPA. Exergames, which integrate MVPA into video game play are an affordable, accessible, home-based exercise program which has shown effectiveness for increasing MVPA and improving both physical and cognitive function in typically developed populations. An exergaming intervention with individual health coaching called GameSquad has been shown to be effective in improving MVPA and cardiometabolic parameters in children with overweight/obesity and adolescents with neurodevelopmental and psychiatric diagnoses. The investigators propose a two phased project to adapt/evaluate the GameSquad intervention for use in adults with DS (GameSquad-DS). In Phase 1, the investigators will utilize a formative approach to develop GameSquad-DS, pilot test the intervention for 4 weeks in 10 young adults with DS and use feedback to refine the intervention for use in Phase 2. In Phase 2, the investigators will conduct a 12-wk. single arm pilot trial in 20 young adults with DS to assess the acceptability, appropriateness, and feasibility of the intervention and calculate effect sizes for change MVPA, physical function, muscular strength, physical activity enjoyment, and self-efficacy. Successful completion of this project represents an initial step in achieving the goal of developing effective interventions to increase MVPA and promote healthy aging in adults with DS.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (18-30 yrs.).
* Diagnosis of DS.
* Sufficient functional ability to understand directions, communicate preferences, wants, and needs through spoken language.
* Living at home with a parent/guardian or in a supported living environment with a parent/caregiver who agrees to serve as a study partner.

Exclusion Criteria:

* Unable to participate in MVPA.
* Serious medical risk, e.g., cancer, recent heart attack, stroke, angioplasty as determined by their primary care provider (PCP).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kirmayer Fitness Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ring-Fit Adventure Group: In Phase 1, participants will be asked to play Ring-Fit Adventure for 60 minutes per week for 4 weeks. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  In Phase 2, participants will be asked to play Ring-Fit Adventure for 60 (wk 1), 90 (wk 2), 120 (wk 3), and 150 (wk 4-12) minutes per week. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  Ring-Fit Adventure Group: Participants will be asked to play the exergame software, Ring-Fit Adventure, and attend weekly virtual health coaching sessions.
Period: Overall Study
Arm/Group | Ring-Fit Adventure Group
Started | 20
Completed | 19
Not Completed | 1
Not completed — One participant ceased contact with the research study team after the initial, pre-testing appt. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (3.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Minutes of Gameplay Per Week
Description: Minutes of Ring-Fit Adventure played per week will be collected from a self-reported sign in sheet.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: minutes/week
Groups:
- Ring-Fit Adventure Group: In Phase 1, participants will be asked to play Ring-Fit Adventure for 60 minutes/week for 4 weeks. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  In Phase 2, participants will be asked to play Ring-Fit Adventure for 60 (wk 1), 90 (wk 2), 120 (wk 3), and 150 (wk 4-12) minutes/week. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  Ring-Fit Adventure Group: Participants will be asked to play the exergame software, Ring-Fit Adventure, and attend weekly virtual health coaching sessions.
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
minutes/week | 100.32 (8.65)

2. Primary Outcome: Retention
Description: Participant retention will be collected.
Time Frame: 12-weeks
Measure: Number; unit: Participants
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 20
Participants | 19

3. Primary Outcome: Attendance
Description: Attendance at 30 min virtual health coaching sessions will be collected.
Time Frame: 12-weeks
Measure: Number; unit: percentage of attended sessions
Units Other Than Participants: health coaching sessions
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
Number analyzed (health coaching sessions) | 228
percentage of attended sessions | 92.45

4. Secondary Outcome: 6-minute Walk Test
Description: This test measures the distance that a participant can walk on a flat, hard surface in a period of 6 minutes. The research team will instruct them on how to prepare and conduct this test.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
Meters
  Pre-Test | 401.13 (92.42)
  Post-Test | 399.26 (81.45)

5. Secondary Outcome: Leg Strength
Description: Leg strength will be measured on the leg press machine. Researchers will assess the maximum amount of weight the participant can press for 5 repetitions.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
Pounds
  Pre-Test | 199.67 (83.34)
  Post-Test | 246.50 (91.61)

6. Secondary Outcome: Hand Grip Strength
Description: The participant will be asked to squeeze a device as hard as they can to test their grip strength. This will be done on both hands.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
Kilograms
  Pre-Testing Left Grip | 20.36 (8.80)
  Post-Testing Left Grip | 19.58 (7.56)
  Pre-Testing Right Grip | 20.15 (8.94)
  Post-Testing Right Grip | 19.72 (7.49)

7. Secondary Outcome: Timed Up and Go
Description: During this test, the participant will be asked to sit down in a chair. Approximately 10 feet in front of the participant there will be a line on the floor. The research team will say "go" and the participant will get up from the chair, walk to the line at a normal pace, and then turnaround and walk back to the chair and sit down again. The research team will record how long it takes to do this.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
Seconds
  Pre-Testing | 6.00 (1.61)
  Post-Testing | 6.14 (1.92)

8. Secondary Outcome: Balance
Description: During this test, the investigators will ask the participant to balance on one leg and reach in three directions as far as they can with their other foot. They will then do the same on the other leg.
Time Frame: 12-weeks
Population: Various participants could not complete certain aspects of the Y-balance test. 3 trials were allowed for each test to ensure testing finished on-time and prevented excess frustration
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
centimeters
  Pre-test anterior reach right leg: number analyzed (Participants) | 12
  Pre-test anterior reach right leg | 48.86 (16.37)
  Post-test anterior reach right leg: number analyzed (Participants) | 12
  Post-test anterior reach right leg | 47.44 (7.57)
  Pre-test anterior reach left leg: number analyzed (Participants) | 12
  Pre-test anterior reach left leg | 47.63 (16.95)
  Post-test anterior reach left leg: number analyzed (Participants) | 12
  Post-test anterior reach left leg | 49.14 (8.02)
  Pre-test posteromedial reach right leg: number analyzed (Participants) | 12
  Pre-test posteromedial reach right leg | 76.03 (17.49)
  Post-test posteromedial reach right leg: number analyzed (Participants) | 12
  Post-test posteromedial reach right leg | 80.75 (12.32)
  Pre-test posteromedial reach left leg: number analyzed (Participants) | 12
  Pre-test posteromedial reach left leg | 76.79 (18.43)
  Post-test posteromedial reach left leg: number analyzed (Participants) | 12
  Post-test posteromedial reach left leg | 80.38 (12.64)
  Pre-test posterolateral reach right leg: number analyzed (Participants) | 8
  Pre-test posterolateral reach right leg | 73.13 (22)
  Post-test posterolateral reach right leg: number analyzed (Participants) | 8
  Post-test posterolateral reach right leg | 73.25 (15.68)
  Pre-Test posterolateral reach left leg: number analyzed (Participants) | 8
  Pre-Test posterolateral reach left leg | 73.13 (17.69)
  Post-Test posterolateral reach left leg: number analyzed (Participants) | 8
  Post-Test posterolateral reach left leg | 70.83 (15.32)

9. Secondary Outcome: Adverse Events
Description: Adverse events will be collected.
Time Frame: 12-weeks
Measure: Number; unit: Adverse Events
Arm/Group | Ring-Fit Adventure Group
Number analyzed (Participants) | 19
Adverse Events | 0

10. Secondary Outcome: Qualitative Interview Data
Description: Semi-Structured interviews will occur after the 12-week intervention to allow participants to make sense of their experience in the intervention.
Time Frame: 12-weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3-months
Description: Intervention safety was defined as the number of participant reports of adverse events. This includes Serious Adverse Events, and Other Adverse Events regardless of whether they were treatment or non-treatment related.
Groups:
- Ring-Fit Adventure Group: In Phase 1, participants will be asked to play Ring-Fit Adventure for 60 minutes per week for 4 weeks. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  In Phase 2, participants will be asked to play Ring-Fit Adventure for 60 (wk 1), 90 (wk 2), 120 (wk 3), and 150 (wk 4-12) minutes per week. Participants will also be asked to attend a weekly, 90 minute health education session with a health educator on zoom.
  Ring-Fit Adventure Group: Participants will be asked to play the exergame software, Ring-Fit Adventure, and attend weekly virtual health coaching sessions.
  No adverse events were reported during the duration of the study.
Arm/Group | Ring-Fit Adventure Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT05473247/Prot_SAP_ICF_000.pdf